CLINICAL TRIAL: NCT03382743
Title: Endocervical Lidocaine Spray for Pain Control During Office Hysteroscopy - a Randomized Control Trial.
Brief Title: Endocervical Lidocaine Spray for Pain Control During Office Hysteroscopy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, sarah mohamed hassan, principal investigator ,lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 171217
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Pain Uterus
Keywords: office hysteroscopy; Lidocaine spray

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Lidocaine group) (Active Comparator): 5 sprays of endocervical Lidocaine 10% spray ( AstraZeneca, bedforshire) are used 3 minutes before office hysteroscopy
  Interventions: Drug: Endocervical Lidocaine spray
- Group B (control group) (No Intervention): office hysteroscopy is done without analgesia

INTERVENTIONS:
Drug: Endocervical Lidocaine spray — 5 sprays of endocervical Lidocaine spray (10%) is used 3 minutes before office hysteroscopy
  Arms: Group A (Lidocaine group)

SUMMARY:
lidocaine spray is used endocervical before office hysteroscopy to reduce the pain

DETAILED DESCRIPTION:
5 sprays of Lidocaine is applied 3 minutes before office hysteroscopy

ELIGIBILITY:
Inclusion Criteria:

Patients indicated for diagnostic hysteroscopy for infertility or AUB. Postmenstrual between days 7 and 11 of the cycle ( except in irregular bleeding)

Exclusion Criteria:

Contraindication to office hysteroscopy Neurological disorders affecting the evaluation of pain. Previous cervical surgery.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Pain sensation | The VAS will be applied immediately after the procedure ended
  The level of pelvic pain will be rated according to a 10-point visual analogue scale (VAS)
Procedure time | immediately after the process
  from introduction of the office hysteroscopy through the external cervical os and the visualization of the uterine cavity

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Kasr El Ainiy Hospital, Cairo
  - Kasr Alaini hospital, Cairo